CLINICAL TRIAL: NCT04363723
Title: The Influence of an Acute Exacerbation During Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease Awaiting Lung Transplantation
Brief Title: The Influence of an Acute Exacerbation During Pulmonary Rehabilitation in COPD Patients Awaiting Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Klaus Kenn (Other)
Collaborators: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Sponsor-Investigator, Klaus Kenn, Professor, Schön Klinik Berchtesgadener Land
Organization: Schön Klinik Berchtesgadener Land (Other)
Other Study IDs: AECOPD pre-LTX
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Exacerbation COPD; pulmonary rehabilitation; lung transplantation; acute exacerbation; waiting list; end-stage lung disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with an acute exacerbation during Rehabilitation: Patients with severe chronic obstructive pulmonary disease awaiting lung Transplantation that developed an acute exacerbation during a pulmonary Rehabilitation program but continued the Rehabilitation program
  Interventions: Other: Pulmonary Rehabilitation
- patients without an acute exacerbation during Rehabilitation: Patients with severe chronic obstructive pulmonary disease awaiting lung Transplantation that did not develop an acute exacerbation during a pulmonary Rehabilitation program and completed the Rehabilitation program regularly.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Patients performed a comprehensive pre-lung transplant inpatient pulmonary rehabilitation program for 4 to 5 weeks duration.

SUMMARY:
Data from chronic obstructive pulmonary disease patients awaiting lung transplantation which performed a pulmonary rehabilitation program will be analyzed retrospectively. Acute exacerbations occur frequently in these patients and have a major impact on the course of the disease. This study investigates the prevalence and the impact of acute exacerbations during pulmonary Rehabilitation in patients with severe chronic obstructive pulmonary disease patients awaiting lung Transplantation that continued the Rehabilitation program despite an acute exacerbation. Data will be taken from the internal database of the reference center (Schoen Klinik Berchtesgadener Land, Schoenau, Germany) where these data were collected during clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of chronic obstructive pulmonary disease including patients with alpha-1 antitrypsin deficiency
* listed for lung Transplantation or in the Evaluation process for lung transplantation
* performed a pulmonary rehabilitation program at the reference center

Exclusion Criteria:

* patients that discontinued the pulmonary Rehabilitation program due to any reason and could therefore not perform assessement tests at the end of regular Rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: data will be collected from the internal database of the reference Center
Sampling Method: Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | day 1 and last day of pulmonary rehabilitation
  The 6-minute walk test will be performed in accordance to the Guidelines of the European Respiratory Society and the American Thoracic Society
Change in Quality of life | day 1 and last day of pulmonary rehabilitation
  health-related Quality of life will be assessed by the physical and mental health component score of the short form 36 health survey (score from 0 to 100 with higher scores indicating better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Rembert A Koczulla, MD, Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

REFERENCES:
- [Derived] Gloeckl R, Jarosch I, Leitl D, Schneeberger T, Nell C, Langer D, Koczulla AR, Kenn K. Influence of an Acute Exacerbation During Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease Awaiting Lung Transplantation. J Cardiopulm Rehabil Prev. 2021 Jul 1;41(4):267-270. doi: 10.1097/HCR.0000000000000613. PMID 34158456